CLINICAL TRIAL: NCT04842084
Title: Determination of Normal Values of Parameters of Thrombin Generation in Fresh PRP and in PPP in Function of Different Tissue Factor Concentrations
Brief Title: Normal Values of Parameters of Thrombin Generation in Function of Different Tissue Factor Concentrations
Acronym: NUAGE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH237; 2021-A00293-38 (Other: ANSM)
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
Keywords: blood; plasma; blood platelets
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy volunteers: Healthy volunteers both sex aged between 18 and 50 without personal or family history of hemorrhage, thrombosis before 45 years old,
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — sampling of 10 S-Monovette tubes (Sarstedt) 4.3 ml of blood specifically for the study representing a total blood volume of 43 ml

SUMMARY:
The thrombin generation assay (TGA) is a good tool for measuring clot formation in plasma.TGA using Calibrated Automated Thrombography method, enables the quantification of thrombin concentrations in platelet-rich plasma (PRP) and in platelet-poor plasma (PPP).According to the clinical context, different TF(Tissue Factor) concentrations (1, 5 and 10 pM) can be used to trigger the coagulation cascade.The aim of the study is to determine the normal values of TG (Thrombin Generation) in fresh PRP and in PPP with different TF concentrations.

DETAILED DESCRIPTION:
The thrombin generation assay (TGA) is a good tool for measuring clot formation in plasma. TGA using Calibrated Automated Thrombography method, enables the quantification of thrombin concentrations in platelet-rich plasma (PRP) and in platelet-poor plasma (PPP). The thrombin generation (TG) profile varies from patient to patient and depends on the activity of the pro and anti-coagulant factors. The TGA values depend on the analytical conditions such as Tissue Factor (TF) concentration and the plasma analyzed (PRP or PPP). According to the clinical context, different TF concentrations (1, 5 and 10 pM) can be used to trigger the coagulation cascade.

As a consequence, the reference values vary with the analytical conditions but also with the studied population (men or women). The reference values are not provided by the manufacturer and each laboratory has to establish the normal values according to the analytical conditions chosen for the pathology explored (hemorrhagic or thrombotic). Moreover, in PPP, the TG results can be different according to batch reagents. That is the reason why plasma will be frozen for a new determination in case of deviation of the result of the control plasma.

The aim of the study is to determine the normal values of TG in fresh PRP and in PPP with different TF concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Patient beneficiary or affiliated to Social security system
* Consent signed

Exclusion Criteria:

* Personal or family history (parents, brothers, sisters) of hemorrhage
* Personal or family history (parents, brothers, sisters) of thrombosis before 45 years old
* Taking an anti-inflammatory or an aspirin one week before the sampling
* Current take of an anticoagulant or antiaggregant treatment
* Surgery within previous month before the sampling
* Chronic pathology responsible of an inflammatory syndrome
* Episode of viral or bacterial infections
* Known HIV or Hepatitis C Virus (HCV) infection
* Participation in a therapeutic clinical trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers both sex aged between 18 and 50 without personal or family history of hemorrhage, thrombosis before 45 years old,
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Thrombin generation parameter in PRP (Peak : nmol thrombin) | At inclusion
  Peak measurement
Thrombin generation parameter in PRP (ETP : nmol*min) | At inclusion
  Endogenous Thrombin Potential measurement
Thrombin generation parameter in PRP (LT : min) | At inclusion
  Lag Time measurement
Thrombin generation parameter in PRP (V : nmol/min) | At inclusion
  Velocity index measurement
Thrombin generation parameter in PRP (TTP : min) | At inclusion
  Time to Peak measurement
Thrombin generation parameter in PRP (ST : min) | At inclusion
  Start Tail measurement

SECONDARY OUTCOMES:
Thrombin generation parameters in PPP (Peak : nmol thrombin) | At inclusion
  Peak measurement
Thrombin generation parameters in PPP (ETP : nmol*min) | At inclusion
  Endogenous Thrombin Potential measurement
Thrombin generation parameters in PPP (LT: min) | At inclusion
  Lag Time measurement
Thrombin generation parameters in PPP (V : nmol/min) | At inclusion
  Velocity index measurement
Thrombin generation parameters in PPP (TTP : min) | At inclusion
  Time to Peak measurement
Thrombin generation parameters in PPP (ST: min) | At inclusion
  Start Tail measurement

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Tardy, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne - Service d'Hématologie, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No